CLINICAL TRIAL: NCT06545188
Title: Impact of Mortality Salience on Treatment Decisions
Acronym: MOST-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: UHN - Princess Margaret Cancer Centre, Toronto, Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GFFU Heigl Foundation 82301
Record Dates: First submitted 2024-07-15; First posted 2024-08-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-02

CONDITIONS: Urological Cancer
Keywords: urological cancer; mortality salience; fear of death; psycho-oncology; decision making; death anxiety
MeSH Terms: conditions — Urologic Neoplasms; Necrophobia

STUDY DESIGN:
Intervention Model Description: Study 1) Urologists: RCT; two arms - Intervention group & control group Study 2) Patients with urological cancer: RCT; two arms - Intervention group & control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mortality salience trigger (Experimental): Mortality Attitudes Personality Survey (MAPS, Rosenblatt et al. 1998) will be administered (two open questions about death and mortality)
  Interventions: Other: Mortality Attitudes Personality Survey
- Dental pain questions (control condition) (Other): Two open questions about a dental treatment will be administered
  Interventions: Other: Dental treatment questions (control condition)

INTERVENTIONS:
Other: Mortality Attitudes Personality Survey — Two open questions about death and mortality will bei administered to trigger mortality salience
  Arms: Mortality salience trigger
Other: Dental treatment questions (control condition) — Two open questions about a dental treatment (control condition)
  Arms: Dental pain questions (control condition)

SUMMARY:
The goal of this clinical trial is to learn if mortality salience has an impact on treatment decisions in urologists and patients with urological cancer. The main questions it aims to answer are:

Does mortality salience lead to more aggressive treatment decisions in a) urologists and b) patients with urological cancer? Which factors predict more aggressive treatment decisions a) in urologists and b) in patients with urological cancer? Is the Fear of cancer recurrence-1 (FCR-1) in German language a valid screening tool for fear of cancer progression in patients with urological cancer?

Researchers will compare a mortality salience trigger to control questions to see if mortality salience leads to more aggressive treatment decisions.

Participants will:

Answer the Mortality Attitudes Personality survey (MAPS) to trigger mortality salience and, in three borderline case vignettes, provide information on how likely they would be to choose a more aggressive therapy.

DETAILED DESCRIPTION:
Background: Harmful overtreatment is a major problem in oncology. Unconscious fear of death (mortality salience) could increase the likelihood of a physician or patient decision in favor of aggressive therapy and thus contribute to overtreatment.

Methods: Conduction of two randomized controlled trials: 1. online survey of n = 260 urological patients, 2. paper questionnaire survey of n = 260 urological cancer inpatients. Intervention group: triggering of mortality salience with two open questions on death, control group: two open questions on dental treatment. The primary endpoint is the probability of opting for aggressive treatment in three questions on a treatment decision Likert scale from 0 to 10). In both studies, the evaluation is carried out as a comparison of means using a two-sided t-test. Secondary endpoints are further factors associated with a decision in favor of aggressive therapy.

Result: An increase in the probability of a decision in favor of the more aggressive therapy as a result of triggering mortality salience is expected with an effect size of d = .35.

Discussion: In order to avoid harmful overtreatment due to unconscious fear of death, doctors could undergo training to deal with their existential fears - this could take place as part of communication training. For cancer patients, this confrontation can take place as part of psycho-oncology training.

ELIGIBILITY:
Study 1) Urologists

Inclusion Criteria:

* sufficient cognitive ability
* German language skills

Exclusion Criteria:

* none

Study 2) Patients

Inclusion Criteria:

* urological cancer (ICD-10: C60, C61, C62, C63, C64, C65, C66, C67, C68)
* age at least 18 years
* German language skills
* sufficient cognitive ability
* capacity to consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
treatment decision | Day 0
  Question about how likely the subject would opt for the more aggressive of two possible therapies on a Likert scale from 0 = very unlikely to 10 = very likely.

SECONDARY OUTCOMES:
Operationalised Psychodynamic Diagnosis (OPD) structure questionnaire, OPD-SQ (Ehrenthal et al., 2015) | Day 0
  12 items, 5-point likert scale, sum score 0 (high level of structure) to 48 (low level of structure) (Ehrenthal et al., 2012)
Relationships-Revised Questionnaire, ECR-RD8 (Ehrenthal et al., 2021) | Day 0
  two subscales: attachment-related avoidance (4 items) and attachment-related anxiety (4 items), 8 items total, 7-point likert scale, sum score from 0 to 48 (higher values correspond to a higher expression of the dimension)
Meaning in Life Questionnaire, MLQ (Steger et al., 2006) | Day 0
  two subscales: search for meaning (5 items) and presence of meaning (5 items), 10 items total, 7-point likert scale, sum score form 5 to 35 per scale with lower levels indicating higher expression of the dimension)
Peace of Mind Scale, POMS (Lee et al., 2013) | Day 0
  7 items, 5-point likert scale, sum score form 7 to 35 (higher levels indicate more peace of mind)
Death Attitude Profile - Revised, DAP-GR | Day 0
  five subscales: fear of death (7 items), death avoidance (5 items), neutral acceptance (5 items), approach acceptance (10 items), escape acceptance (5 items), 35 items total, 7-point likert scale, an average value is calculated for each subscale by dividing the sum score of the domain by the number of its items
Urologists - socio-demographics | Day 0
  age (years), gender (male, female, other), relationship status (yes, no), children (yes, no), underage children living in the same household (yes, no)
Urologists - job related factors | Day 0
  professional experience (years), position (chief physician, senior physician, specialist, assistant physician), place of work (hospital, practice, both, other)
Urologists - Effort-Reward-Imbalance Questionnaire - short version, ERI (short version) (Siegrist et al., 2009) | Day 0
  Three subscales: Effort (7 items), reward (3 items), work stress (6 items), 16 items total, 4-point-likert scale (1 to 4), sum scores for each domain with higher levels corresponding to higher expression of the dimension
Patients - (modified) psycho-oncological basic documentation, PO-Bado (Herschbach et al., 2004) | Day 0
  gender (male, female, other), partnership (yes, no) children (yes, no), underage children living in the same household (yes, no), work situation (employed, on sick leave, housework, pension, unemployed, other [free text]), metastases (yes, no, unknown), date of first diagnosis (month/year, unknown), current disease status (first disease, second disease, relapse, remission, unknown), treatments in the last two months (surgery, radiation, chemotherapy, other systemic therapy / drug treatment for cancer (e.g. immunotherapy), hormones, none, other [free text]), other relevant physical illnesses (yes, which? Immunotherapy), hormones, none, other [free text]), other relevant physical illnesses (yes, which? [free text], no, not known), psychotropic drugs / opiates (yes, which? [free text], no, not known), psychological / psychiatric treatment in the past? (yes, no, not known)
Patients - socio-demographics | Day 0
  age (years), education (no school-leaving certificate, primary school leaving certificate, secondary school leaving certificate ('Hauptschule' or 'Realschule'), Polytechnical high school 10th grade (before 1965: 8th grade), technical secondary school leaving certificate, high school diploma, I have another school-leaving certificate, namely: [free text])
Patients - European Health Literacy Survey 16, HLS-EU-Q16 (Röthlin et al., 2013) | Day 0
  Four dimensions: accessing, understanding, assessing and using health information, 16 items, four response categories are binarized (1 = "very easy / "fairly easy"; 0 = "very difficult" / "fairly difficult") and added together to form a total score: "adequate" (13-16 points), "problematic" (9-12 points) and "inadequate" (1-8 points).
Patients - Patient Health Questionnaire 9, PHQ-9 (Kroenke et al., 2001) | Day 0
  A total score (0 - 27 points) is calculated from nine items on a four-point Likert scale. The following grading can be used: 0 - 4 points: minimal depressive symptoms, 5 - 9 points: mild depressive symptoms, 10 - 14 points: mild depressive symptoms, 15 - 19 points: moderate depressive symptoms, 20 - 27 points: severe depressive symptoms.
Patients - Generalized Anxiety Disorder 7, GAD-7 (Löwe et al., 2008) | Day 0
  A total score (0 - 21 points) is calculated from seven items, each with a four-point Likert scale. The threshold value for increased anxiety is 10 points.
Patients - Short form of the Fear of Progression Questionnaire (FoP-Q-SF) (Mehnert et al., 2006) | Day 0
  The questionnaire comprises 12 items with a five-point Likert scale, from which a total score of 12 to 60 points can be calculated. Moderate progressive anxiety is present if more than 50 % of the questions are answered with "often" or "very often", high progressive anxiety with more than 75 % of the questions.
Patients - fear of cancer recurrence | Day 0
  Fear of cancer recurrence, FCR-1r (Smith et al., 2023)
  1 item, scale from 0 (no fear of recuurence) to 10 (high fear of recurrence)
Patients - Concerns about Recurrence Questionnaire-4, CARQ-4 (Thewes et al. 2015) | Day 0
  The first three items are rated on an 11-point Likert scale from 0 to 10. Item 4 asks for the subjective probability of cancer recurrence (0 to 100), which is then converted to a 0-10 scale. Thus, the total score ranges from 0 to 40, with scores of 12 or higher indicating elevated fear of cancer recurrence levels.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Fugmann, Dr. med., Principal Investigator — Heinrich Heine University Duesseldorf, Germany
Locations (1):
- University Hospital Düsseldorf, Department of Urology, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No